CLINICAL TRIAL: NCT01744249
Title: A Phase II/III Randomized Double-blind Study of Sandostatin LAR in Combination With Axitinib Versus Sandostatin LAR With Placebo in Patients With Advanced G1-G2 Neuroendocrine Tumours (WHO 2010) of Non-pancreatic Origin
Brief Title: Sandostatin LAR and Axitinib vs Pbo in Pnts With Advanced Well-differentiated Non-pancreatic Neuroendocrine Carcinomas
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXI-IIG-02; 2011-001550-29 (EudraCT Number)
Record Dates: First submitted 2012-09-25; First posted 2012-12-06 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Neuroendocrine Tumors; Advanced Cancer
Keywords: Advanced neuroendocrine tumours of non-pancreatic origin; axitinib
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axitinib + Sandostatin LAR (Experimental): Axitinib 5 mg BID + Sandostatin LAR 30mg/28 days
  Interventions: Drug: Axitinib; Drug: Sandostatin LAR
- Placebo + Sandostatin LAR (Placebo Comparator): Placebo BID + Sandostatin LAR 30mg/28 days
  Interventions: Drug: Sandostatin LAR; Drug: Placebo

INTERVENTIONS:
Drug: Axitinib — Orally, 5mg, twice daily, until progression or until unacceptable toxicity, with or without food intake.
  Arms: Axitinib + Sandostatin LAR
Drug: Sandostatin LAR — Intramuscular, 30mg, single injection every 28 days, until disease progression or unacceptable toxicity
Drug: Placebo — orally, twice daily, until disease progression or unacceptable toxicity, with or without food intake.
  Arms: Placebo + Sandostatin LAR

SUMMARY:
Assess whether therapy with axitinib, a potent angiogenic inhibitor of the tyrosine kinase receptors of VEGF bioavailable by oral administration, is capable of improving PFS in patients with advanced G1-G2 NETs of nonpancreatic origin with progressive disease documented in the 12 months prior to entering the study.

DETAILED DESCRIPTION:
Phase II/III, prospective, multicenter, randomized (1:1), double-blind study to evaluate the efficacy and tolerability of axitinib in patients diagnosed with advanced G1-G2 neuroendocrine tumors (WHO 2010) of nonpancreatic origin that have presented documented disease progression in the 12 months prior to entering the study. In the first part of the study (Phase II), 105 patients were enrolled. The second part of the study is the expansion to Phase III, which is expected to include 148 additional patients. Patients will be randomized to receive Sandostatin LAR with axitinib or Sandostatin LAR with placebo until disease progression or unacceptable toxicity occurs. Randomization will be stratified by the time from diagnosis to enrollment in the study (more vs less than or equal to 12 months), the origin of the primary tumor (gastrointestinal tract vs non-gastrointestinal tract [lung or other sites]) and ki-67 (< 5% vs > 5%).

ELIGIBILITY:
Inclusion Criteria:

1. G1-G2 neuroendocrine tumor (WHO 2010) of histologically confirmed non-pancreatic origin, functioning and nonfunctioning
2. Metastatic or locally advanced disease not amenable to treatment with curative intent
3. Clinical and/or radiological disease progression documented in the 12 months prior to study entry.
4. Patients should have at least one measurable lesion as defined by RECIST 1.1 criteria. Patients should not have undergone local or regional ablative procedures (embolization, cryoablation, radiofrequency ablation, or others) in the 6 months prior to entering the study, unless there are other locations of measurable disease or clear radiological progression after carrying out these procedures (in these cases, local and regional ablation procedures shall be permitted if they have been performed at least 1 month prior to enrollment in the study).
5. Ki-67 < 20%
6. Prior treatment with somatostatin analogues is allowed
7. Prior treatment with interferon is allowed
8. Prior treatment is allowed with up to 2 antineoplastic systemic treatment lines different from SAs or IFN (systemic treatment is understood as conventional cytotoxic chemotherapy or new drugs for therapeutic targets as mTOR or other, as long as it is not directed against VEGF/VEGFR). Treatment with SAs or IFN does not count as prior lines of antineoplastic treatment.
9. Prior treatment with targeted therapy against VEGF or VEGFR is not allowed.
10. Adequate organ function as defined by the following criteria:

    * Absolute neutrophil count ≥ 1500 cells/mm3,
    * Platelet count ≥ 75,000 cells/mm3,
    * Hemoglobin ≥ 9.0 g/dL,
    * AST y ALT ≤ 2.5 x upper limit of normal (ULN), except if liver metastases exist, in which case AST and ALT 5.0 ≤ x ULN is allowed,
    * Total bilirubin ≤ 1.5 x ULN,
    * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min,
    * Proteinuria < 2+ by reactive strip. If the reactive strip is ≥ 2+, a 24-hour urine sample should be collected and the patient may be eligible if urinary protein excretion is < 2 g every 24 hours.
11. Men or women aged ≥ 18 years.
12. ECOG performance status 0-2
13. Life expectancy ≥ 12 weeks
14. At least 4 weeks should pass from the end of the previous systemic treatment with resolution of all treatment-related toxicities to grade ≤ 1 according to NCI CTCAE Version 4.0 or to baseline, except for alopecia or properly treated hypothyroidism.
15. No prior evidence of uncontrolled hypertension should exist, as documented by 2 baseline blood pressure readings taken at least 1 hour apart. Baseline readings of systolic blood pressure should be ≤ 150 mm Hg and baseline readings of diastolic pressure should be ≤ 90 mm Hg. Patients whose hypertension is being controlled with antihypertensive therapy are eligible.
16. Women (or their partners) should be surgically sterilized or postmenopausal, or must agree to use an effective contraceptive method during and for at least 6 months after receiving study treatment. All women of childbearing age should have a negative pregnancy test (serum/urine) within 7 days prior to starting treatment. Men (or their partners) should be surgically sterilized or must agree to use an effective contraceptive method during and for at least 6 months after receiving study treatment. The definition of an effective contraceptive method must comply with local regulations and will be based on the criterion of the principal investigator or a designated associate. Lactating women may not participate in this study.
17. Signed and dated informed consent document stating that the patient has been informed of all the pertinent aspects of the trial prior to recruitment.
18. Willingness and ability to comply with scheduled visits, treatment plans (including willingness to take axitinib or placebo according to randomization), laboratory tests, and other study procedures.

Exclusion Criteria:

1. Subjects must be evaluated with regard to the following exclusion criteria:

1. The following types of endocrine tumors will not be included: paraganglioma, adrenal endocrine tumor, thyroid, parathyroid, or pituitary.
2. Major surgery within previous 4 weeks, or radiation therapy within 2 weeks prior to the start of treatment. Prior palliative radiotherapy for metastatic lesions is permitted if there is at least one measurable lesion that has not been irradiated (i.e., if there are other non-irradiated target lesions).
3. Gastrointestinal abnormalities, including:

   * Inability to swallow oral medication;
   * Need for intravenous feeding;
   * Prior surgical procedures that affect absorption, including total gastric resection;
   * Treatment for active peptic ulcer in the last 6 months;
   * Uncontrolled active gastrointestinal bleeding unrelated to cancer, as evidenced by hematemesis, hematochezia or clinically significant melena in the last 3 months without evidence of resolution documented by endoscopy or colonoscopy;
   * Malabsorption syndromes;
4. Current or anticipated need for treatment with drugs that are potent inhibitors of CYP3A4 (grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, and delavirdine) unless they can be replaced by another medication with minimal potential for CYP3A4/5 inhibition. The use of low-dose oral steroids (< 5 mg/day prednisone or equivalent) is allowed. Co-administration of steroids may increase plasma concentrations of axitinib.
5. Current use or anticipated need for treatment with drugs that are known potent CYP3A4/5 inducers (carbamazepine, dexamethasone, felbamate, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampicin, and St. John's wort) unless they can be replaced by another medication with minimal potential for CYP3A4 induction. Co-administration of CYP3A4/5 inducers may decrease plasma concentrations of axitinib.
6. Need for anticoagulant therapy with oral vitamin K antagonists. Low doses of anticoagulants to maintain the patency of a central venous access device or to prevent deep vein thrombosis are permitted. Use with therapeutic doses of low molecular weight heparin is allowed.
7. Clinically relevant history of bleeding in the last 6 months, including severe hemoptysis or hematuria, unless it has been due to a treated cause (e.g., completely resected bleeding intestinal tumor).
8. Active epilepsy or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
9. Serious uncontrolled illness or active infections that may interfere with the patient's ability to receive the study treatment.
10. Any of the following events in the 12 months prior to administration of the study drug: myocardial infarction, uncontrolled angina, implantation of a coronary or peripheral bypass, symptomatic congestive heart failure, stroke or transient ischemic attack. Deep vein thrombosis or pulmonary embolism in the prior 6 months.
11. Ongoing grade ≥ 2 cardiac arrhythmias according to NCI CTCAE: atrial fibrillation of any grade or QTc interval > 450 ms for men or > 470 ms for women.
12. Patients with human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome-related disease.
13. Prior history of cancer except those treated with curative intent for non-melanoma skin cancer in situ, breast or cervical cancer in situ, or those treated for any cancer with curative intent and no evidence of disease in the last 5 years prior to enrollment in the study.
14. Dementia or significantly altered mental status that could prevent compression, or submission of informed consent and compliance with the requirements of this protocol.
15. Any severe, acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with participation in the study or with study drug administration, or that may interfere with the interpretation of results, and that could interfere with the patient's ability to take part in this study in the investigator's opinion.
16. The patient's participation or intention to participate (in the 4 weeks prior to starting drug administration) in a study in which the patient will receive an investigational medicinal product.
17. Subjects who are institutionalized by governmental or by judicial decision, or subjects who are dependent of the sponsor, the investigator or the trial site will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2011-11 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of axitinib in terms of PFS | until disease progression, end of treatment or minimum 6 months
  calculated from the date of random assignment until the date of first progressive disease or tumor-related death

SECONDARY OUTCOMES:
Objective response rate (ORR) and the duration of response. | Until disease progression, end of treatment or minimum 6 months
  Measured according to RECIST 1.1 criteria; Sum of longest diameter of target lesions measured in mm
Functional response rate using F-DOPA-PET (optional, depending on availability) | Until disease progression, end of treatment or minimum 6 months
  measured in SUV (standardized uptake value)
Biochemical response (5-OH-indoleacetic acid and chromogranin A) | Until death, last follow-up, or minimum 6 months
  measurable in mL/ 24h and ng/ml respectively, through blood and urine test
Safety and tolerability of axitinib (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE], version 4.0) | Until disease progression, end of treatment or minimum 6 months
  All adverse events and serious adverse events will be monitored with regular monitoring of hematology and blood chemistry parameters and regular physical examinations. Adverse events will be evaluated continuously throughout the study. Safety and tolerability will be assessed according to the National Institute of Health/National Cancer Institute (NIH/NCI) Common Terminology Criteria for Adverse Events version 4 (CTCAE v4)
Explore potential biomarkers | Until disease progression or or minimum 6 months
  The following parameters will be measured: circulating tumor cells, circulating endothelial cells, hypertension (mmHg), and other serum or tumoral biomarkers of angiogenesis).
  Peripheral blood samples (9ml) will be obtained before treatment, after 1 month since the start of treatment and after disease progression and or the end of study visit. The blood samples will be processed for mRNA extraction. Hypoxia dependant genes and marker genes which transcription depends on the activation of VEGF, will be analyzed using qPCR. The dynamic profile of those genes will then be analyzed in relation to the response to axitinib, evaluating their predictive value of response.
  Paraffin-embedded tumor tissue will also be collected from all patients to investigate the prognostic value and predictive potential of the different intracellular pathways related to VEGFR, PDGFR and other signaling pathways.
Evaluate overall survival. | from the date of randomization to the date of death from any cause whichever came first, assessed up to 50 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Garcia Carbonero, MD, Study Chair — Hospital 12 de Octubre
Locations (26):
- Marburg Universitätsklinikum Giessen und Marburg GmbH, Marburg, Germany
- Italy (2):
  - Azienda Ospedaliera Universitaria di Perugia, Perugia
  - Sapienza, Universitá di Roma, Ospedale sant'Andrea, Rome
- Spain (22):
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Hospitalario Univ A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Virgen de las Nieves, Granada
  - Hospital universitario de Leon, León
  - MD Anderson Cancer Center, Madrid
  - Hospital Clara Campal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Univ La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Univ de Salamanca, Salamanca
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Clatterbridge Cancer Centre, Bebington, Wirral, United Kingdom

REFERENCES:
- [Derived] Kunz PL. Angiogenesis inhibitors in neuroendocrine tumours: finally coming of age. Lancet Oncol. 2020 Nov;21(11):1395-1397. doi: 10.1016/S1470-2045(20)30560-X. No abstract available. PMID 33152282